CLINICAL TRIAL: NCT01890005
Title: Low Dose Aspirin Between 13 and 16 Weeks of Pregnancy for the Prevention of Preeclampsia. Double Blind, Randomized, Controlled Trial.
Brief Title: Low Dose Aspirin for the Prevention of Preeclampsia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MHST2013-05
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Low dose aspirin; Fetal growth restriction; Neonatal death; Stillbirth; Abruptio placenta
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Perinatal Death; Stillbirth; Abruptio Placentae | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Experimental): Low dose aspirin (100 mg) starting between 13 and 16 weeks of pregnancy until 36 weeks of pregnancy, taken at night.
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo (identical to low dose aspirin (100 mg)) starting between 13 and 16 weeks of pregnancy until 36 weeks of pregnancy, taken at night.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Low dose aspirin (100 mg) starting between 13 and 16 weeks of pregnancy until 36 weeks of pregnancy, taken at night.
  Arms: Aspirin
Drug: Placebo — Placebo starting between 13 and 16 weeks of pregnancy until 36 weeks of pregnancy, taken at night.
  Arms: Placebo

SUMMARY:
Preeclampsia is one of the three leading causes of maternal morbidity and mortality all over the world. The use of low dose aspirin has been mentioned in several studies with promising results. The investigators decided to evaluate the use of low dose aspirin, starting between 13 and 16 weeks of pregnancy, based on clinical characteristics only to reduce the incidence of preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 13 and 16 weeks of pregnancy
* High risk of preeclampsia, based in clinical risk factors as:

Preeclampsia in a previous pregnancy Mother or sister that developed preeclampsia in a previous pregnancy Diabetes Mellitus (insulin dependant) Chronic Hypertension (with/without proteinuria) Body Mass Index > 32 Multiple pregnancy Lupus or other autoimmune disorder Chronic Renal Disease.

Exclusion Criteria:

* Blood coagulation disorders of any kind
* Peptic ulcers
* Allergy to aspirin
* Chronic use of anti-inflammatory drugs
* Fetus with mayor anomalies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Prevention of preeclampsia | 6 months
  The number of cases of preeclampsia that appear in both groups before 34 weeks of pregnancy

SECONDARY OUTCOMES:
Prevention of preeclampsia at term | 6 months
  The number of cases of preeclampsia that appear in both groups between 37 and 41 weeks of pregnancy.
Stillbirth | 6 months
  The number of cases of stillbirths that appear in both groups at any given time during pregnancy.
Neonatal deaths | 6 months
  The number of cases of neonatal deaths that appear in both groups, regardless of the cause.
Neonatal intensive care unit admissions. | 28 days
  The number of cases that require admittance to the Neonatal Intensive Care Unit in both groups in the first 28 days after birth.
Abruptio placenta | 6 months
  The number of cases of abruptio placenta that appear in both groups at any given time during pregnancy.
Fetal Growth Restriction | 6 months
  The number of cases of fetal growth restriction, defined as a fetal weight below the 10th percentile and an abnormal umbilical cord doppler that appear in both groups at any given time during pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Principal Investigator — Saint Thomas Maternity Hospital; Rodrigo Velardee, MD, Principal Investigator — Saint Thomas Maternity Hospital; Ameth Hawkins, MD, Principal Investigator — Saint Thomas Maternity Hospital; Ana Moreno, MD, Principal Investigator — Saint Thomas Maternity Hospital
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Panama